CLINICAL TRIAL: NCT02773524
Title: A Randomised Phase III Double-Blind Placebo-Controlled Study of Regorafenib in Refractory Advanced Gastro-Oesophageal Cancer (AGOC)
Brief Title: A Study of Regorafenib in Refractory Advanced Gastro-Oesophageal Cancer
Acronym: INTEGRATEIIa
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Collaborators: Canadian Cancer Trials Group (Network); Academic and Community Cancer Research United (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG0315OG
Record Dates: First submitted 2016-05-04; First posted 2016-05-16 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Gastro-Oesophageal Cancer
Keywords: Metastatic; Locally recurrent; Oesophago-gastric junction; Stomach; Adenocarcinoma; Undifferentiated Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Adenocarcinoma; Carcinoma | interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Regorafenib (Experimental): Regorafenib 160mg (4 x 40 mg tablets) orally, once daily on days 1-21 of each 28 day cycle + best supportive care until progression
  Interventions: Drug: Regorafenib
- Placebo (Placebo Comparator): Placebo 160mg (4 x 40 mg tablets) orally, once daily on days 1-21 of each 28 day cycle + best supportive care until progression
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Regorafenib — Regorafenib is the experimental intervention in this study. Regorafenib will be self-administered by participants at 160mg (4 x 40mg tablets) orally once daily on days 1-21 of each 28 day cycle plus best supportive care until progression or prohibitive toxicity as defined by the protocol.
  Other Names: Stivarga
  Arms: Regorafenib
Other: Placebo — Placebo (matching in appearance to regorafenib) made of microcrystalline cellulose, will be self-administered by participants at 160mg (4 x 40mg tablets) orally once daily on days 1-21 of each 28 day cycle plus best supportive care until progression or prohibitive toxicity as defined by the protocol.
  Arms: Placebo

SUMMARY:
A randomised phase III, double-blind, placebo-controlled trial with 2:1 (regorafenib : placebo)

DETAILED DESCRIPTION:
Purpose:

The purpose of this Phase III study is to determine if regorafenib improves overall survival in patients with Advanced Gastro-Oesophageal Carcinoma.

Who is it for:

You may be eligible to join this study if you are aged 18 years or above and have been diagnosed with advanced (metastatic or locally recurrent) Gastro-Oesophageal Carcinoma which has not responded to a minimum of 2 lines of prior anti-cancer therapy.

Trial Details:

Participants will be randomly (by chance) allocated to one of two groups: regorafenib or placebo in 2:1 ratio respectively and will not be aware of their group allocation. Regorafenib or matching placebo will be self-administered by participants orally once daily on days 1-21 of each 28 days cycle. Treatment will continue until disease progression or prohibitive toxicity. Participants will be followed up every 2-4 weeks in order to evaluate their progress on the study.

ELIGIBILITY:
Inclusion Criteria

1. Adults (18 years or over) with metastatic or locally recurrent gastro-oesophageal cancer which:

   1. has arisen in any primary gastro-oesophageal site (oesophago-gastric junction (GOJ) or stomach); and
   2. is of adenocarcinoma or undifferentiated carcinoma histology , and
   3. is evaluable according to Response Evaluation Criteria in Solid Tumours (RECIST Version 1.1) by computed tomography (CT) scan performed within 21 days prior to randomisation. A lesion in a previously irradiated area is eligible to be considered as measurable disease as long as there is objective evidence of progression of the lesion prior to study enrolment; and
   4. has failed or been intolerant to a minimum of 2 lines of prior anti-cancer therapy for recurrent/metastatic disease which must have included at least one platinum agent and one fluoropyrimidine analogue.

      Note: Neoadjuvant or adjuvant chemotherapy or chemoradiotherapy will be considered as first line treatment where people have relapsed or progressed within 6 months of completing treatment; Radiosensitising chemotherapy given solely for this purpose concurrent with palliative radiation will not be considered as a line of treatment. Ramucirumab monotherapy, or immunotherapy with a checkpoint inhibitor, will be considered a line of treatment.
   5. HER2-positive participants must have received trastuzumab.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
3. Ability to swallow oral medication.
4. Adequate bone marrow function (Platelets ≥100x109/L; Absolute Neutrophil Count (ANC) ≥1.5x109/L and Haemoglobin ≥ 9.0g/dL).
5. Adequate renal function (Creatinine clearance >50 ml/min) based on either the Cockcroft-Gault formula (Appendix 2), 24-hour urine or Glomerular Filtration Rate (GFR) scan; and serum creatinine ≤1.5 x Upper Limit of Normal (ULN).
6. Adequate liver function (Serum total bilirubin ≤1.5 x ULN, and INR ≤ 1.5 x ULN, and Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase (ALP) ≤2.5 x ULN (≤ 5 x ULN for participants with liver metastases)). Participants being treated with an anti-coagulant, such as warfarin or heparin, will be allowed to participate provided that no prior evidence of an underlying abnormality in these parameters exists.
7. Adequate cardiac function (Left Ventricular Ejection Fraction (LVEF) ≥ 50% or above the lower limit of normal (LLN) for the Institution (whichever is lower). Cardiac function should be assessed within 3 months prior to randomisation, but after completion of any anthracycline-containing chemotherapy.
8. Willing and able to comply with all study requirements, including treatment, timing, and/or nature of required assessments and follow-up.
9. Study treatment both planned and able to start within 7 days after randomisation (note: subjects randomised on a Friday should commence treatment no earlier than the following Monday).
10. Signed, written informed consent.

Exclusion Criteria

1. Known allergy to the investigational product drug class or excipients in the regorafenib.
2. Poorly-controlled hypertension (systolic blood pressure >140mmHg or diastolic pressure> 90mmHg despite optimal medical management).
3. Participants with known, uncontrolled malabsorption syndromes.
4. Any prior anti-VEGF targeted therapy using small molecule VEGF TKIs (e.g. apatinib). Prior anti-VEGF targeted monoclonal antibody therapies (e.g. bevacizumab and ramucirumab) are permitted.
5. Treatment with any previous drug therapy within 2 weeks prior to first dose of study treatment. This includes any investigational therapy.
6. Use of biological response modifiers, such as granulocyte colony stimulating factor (G-CSF), within 3 weeks prior to randomisation.
7. Concurrent treatment with strong CYP3A4 inhibitors or inducers.
8. Palliative radiotherapy, unless more than 14 days have elapsed between completion of radiation and the date of registration, and adverse events resulting from radiation have resolved to< Grade 2 according to CTCAE V4.03.
9. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization.
10. Arterial thrombotic or ischaemic events, such as cerebrovascular accident, within 6 months prior to randomization.
11. Venous thrombotic events and pulmonary embolism within 3 months prior to randomization.
12. Any haemorrhage or bleeding event ≥ Grade 3 according to CTCAE v4.03 within 4 weeks prior to randomization.
13. Non-healing wound, ulcer, or bone fracture.
14. Interstitial lung disease with ongoing signs and symptoms.
15. Clinical hyperthyroidism or hypothyroidism. Note: non-clinically significant abnormal TFTs (abnormal TSH and abnormal T3 and/or abnormal T4) considered to be due to sick euthyroid syndrome is allowed.
16. Persistent proteinuria of ≥ Grade 3 according to CTCAE v4.03 (equivalent to > 3.5g of protein over 24 hours, measured on either a random specimen or 24 hour collection).
17. Uncontrolled metastatic disease to the central nervous system. To be eligible, CNS metastases should have been treated with surgery and/or radiotherapy and the patient should have been receiving a stable dose of steroids for at least 2 weeks prior to randomization, with no deterioration in neurological symptoms during this time.
18. History of another malignancy within 2 years prior to randomization. Participants with the following are eligible for this study:

    1. curatively treated cervical carcinoma in situ,
    2. non-melanomatous carcinoma of the skin,
    3. superficial bladder tumours (T1a [Non-invasive tumour], and Tis[Carcinoma in situ]),
    4. treated thyroid papillary cancer
19. Any significant active infection, including chronic active hepatitis B, hepatitis C, or HIV. Testing for these is not mandatory unless clinically indicated. Participants with known Hepatitis B/C infection will be allowed to participate providing evidence of viral suppression has been documented and the patient remains on appropriate anti-viral therapy.
20. Serious medical or psychiatric condition(s) that might limit the ability of the patient to comply with the protocol.
21. Pregnancy, lactation, or inadequate contraception. Women must be post-menopausal infertile, or use a reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to randomization. Men must have been surgically sterilized or use a barrier method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From time of patient randomisation until date last known alive (up to 12 months following end of treatment).
  The interval from the date of randomisation to date of death from any cause, or the date last known alive.

SECONDARY OUTCOMES:
Progression Free Survival | From time of patient randomisation until first evidence of disease progression or death (up to 12 months following randomisation).
  The interval from the date of randomisation to the date of first evidence of disease progression or death, whichever occurs first.
Objective Tumour Response Rate | From time of patient randomisation until evidence of complete or partial response (up to 12 months following randomisation).
  The OTRR will be calculated by summing the number of participants in a given arm that are assessed as having a complete or partial response (as per RECIST criteria), and dividing this by the total number of participants in the corresponding arm of the analysis set.
Evaluation of health states experienced by participants | From time of commencement of treatment until first evidence of disease progression (up to 12 months following commencement of treatment).
  Questionnaire used to assess quality of life
Rates of Adverse Events | From time dose of study treatment until 30 days after last dose of study treatment
  A descriptive analysis of the adverse events (AE) data will be prepared for participants in the safety population. The number and percentage of participants who experience AEs will be tabulated according to CTCAE term/category, grade, and seriousness.

OTHER OUTCOMES:
Identification of tumour markers to that predict treatment outcomes for AGOC | Up to 24 months following close of recruitment.
  Biomarker assessment, CTC DNA assessment to predict whether treatment for AGOC is efficacious
Evaluation of regorafenib Maximum Plasma Concentration [Cmax] between Asia and Rest of World cohorts. | Up to 24 months following close of recruitment.
  Evaluation of regorafenib Maximum Plasma Concentration [Cmax] in patients from either Asia or ROW to assess whether genetic factors aide/hinder metabolic rate of consumption of regorafenib

CONTACTS AND LOCATIONS:
Overall Officials: Nick Pavlakis, Prof, Study Chair — AGITG
Locations (60):
- United States (4):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - USC Norris, Los Angeles, California
  - Carle Cancer Center NCI Community Oncology Research Program, Urbana, Illinois
  - Bon Secours Cancer Institute, Midlothian, Virginia
- Australia (26):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Border Medical Oncology, Albury, New South Wales
  - Monash Medical Centre, Clayton, New South Wales
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St Vincent's Public Hospital, Darlinghurst, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Newcastle Private Hospital, New Lambton Heights, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Ballarat Oncology and Haematology Services, Wendouree, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Darwin Hospital, Tiwi, Northern Territory
  - The Townsville Hospital, Douglas, Queensland
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Sunshine Coast University Hospital, Sunshine Coast, Queensland
  - Ashford Cancer Centre Research, Ashford, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Austin Hospital, Heidelberg, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - St John of God Hospital Subiaco, Subiaco, Western Australia
- Canada (7):
  - PEI Cancer Treatment Centre, Queen Elizabeth Hospital, Charlottetown
  - Queen Elizabeth II Health Sciences Centre, Nova Scotia
  - Ottawa Hospital Research Institute, Ottawa
  - The Research Institute of the McGill University Health Centre, Québec
  - Allan Blair Cancer Centre, Regina
  - Saskatoon Cancer Centre, Saskatoon
  - University Health Network Princess Margaret Cancer Centre, Toronto
- Japan (2):
  - National Cancer Centre Hospital East, Chiba, Kashiwa
  - Hokkaido University Hospital, Sapporo, Kita
- Auckland Hospital, Auckland, New Zealand
- South Korea (15):
  - Hallym University Sacred Heart Hospital, Anyang
  - Dong-A University Hospital, Busan
  - Chonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Chung-Ang University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea - Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea - Yeouido St. Mary's Hospital, Seoul
  - Yonsei University Health System - Gangnam Severance Hospital, Seoul
  - Yonsei University Health System - Severance Hospital, Seoul
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Taipei
  - National Taiwan University Hospital (NTUH), Taipei
  - Taipei Veterans General Hospital (TPVGH), Taipei

REFERENCES:
- [Derived] Soon YY, Sjoquist K, Marschner IC, Schou IM, Pavlakis N, Goldstein D, Shitara K, Stockler MR, Simes J, Martin AJ. INTEGRATE pooled phase 2/3 results are robust to postprogression switching and the winner's curse. JNCI Cancer Spectr. 2025 Jul 1;9(4):pkaf053. doi: 10.1093/jncics/pkaf053. PMID 40455046
- [Derived] Pavlakis N, Shitara K, Sjoquist K, Martin A, Jaworski A, Tebbutt N, Bang YJ, Alcindor T, O'Callaghan C, Strickland A, Rha SY, Lee KW, Kim JS, Bai LY, Hara H, Oh DY, Yip S, Zalcberg J, Price T, Simes J, Goldstein D. INTEGRATE IIa Phase III Study: Regorafenib for Refractory Advanced Gastric Cancer. J Clin Oncol. 2025 Feb;43(4):453-463. doi: 10.1200/JCO.24.00055. Epub 2024 Oct 4. PMID 39365958
- [Derived] Lam LL, Pavlakis N, Shitara K, Sjoquist KM, Martin AJ, Yip S, Kang YK, Bang YJ, Chen LT, Moehler M, Bekaii-Saab T, Alcindor T, O'Callaghan CJ, Tebbutt NC, Hague W, Chan H, Rha SY, Lee KW, Gebski V, Jaworski A, Zalcberg J, Price T, Simes J, Goldstein D. INTEGRATE II: randomised phase III controlled trials of regorafenib containing regimens versus standard of care in refractory Advanced Gastro-Oesophageal Cancer (AGOC): a study by the Australasian Gastro-Intestinal Trials Group (AGITG). BMC Cancer. 2023 Feb 22;23(1):180. doi: 10.1186/s12885-023-10642-7. PMID 36814222